CLINICAL TRIAL: NCT00156312
Title: Evaluation of Thymidine Phosphorylase and Other Predictive/Prognostic Factors in Primary Breast Cancer Treated With Docetaxel and Capecitabine (DC)
Brief Title: Evaluation of Tumor Factors in Breast Cancer Treated With Docetaxel and Capecitabine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: The cancer answer line, U of M
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: UMCC 2003.045
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel
Drug: Capecitabine

SUMMARY:
The purpose of this study is to determine whether the combination of the drugs docetaxel and capecitabine is effective in treating breast cancer patients.

DETAILED DESCRIPTION:
Some chemotherapy drugs are thought to work in synergy, meaning they work better in combination, rather than singly because one drug may cause changes in the tumor that will make the other drug more effective. The drugs docetaxel and capecitabine may work in synergy, based on laboratory studies in tumors. These laboratory studies show that docetaxel increases the levels of a critical enzyme, called thymidine phosphorylase (TP), which is necessary to activate the capecitabine. This study will use this promising chemotherapy combination in patients with breast cancer. Before, during, and after chemotherapy, the participants' breast tumors will be examined to see if TP increases, as predicted by the laboratory studies. The study will also look at other factors in tumors and blood that may be able to predict how effective the chemotherapy will be for each individual, so that in the future we may better select the best chemotherapy for an individual's cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a primary measurable invasive breast cancer with the primary tumor intact (T1, 2, 3, or 4, any N, M0). The clinical stage must meet one of the following criteria:

  1. Size ≥ 2 cm on mammography, ultrasound, or PE
  2. OR ≥ 1 cm and ER negative, and amenable to research biopsy.
  3. OR <1 cm and documented intact axillary metastasis amenable to serial research CORE biopsies.
* Histologic diagnosis of at least one site of invasive cancer must be by core needle biopsy or incisional biopsy. Immunohistochemical staining for estrogen and progesterone receptors, and HER-2 neu receptor should be obtained on the initial diagnostic sample.
* Patients must have had mammography performed at the University of Michigan, OR outside film review prior to enrollment.
* Patients must have clinical ultrasound performed at the University of Michigan prior to enrollment.
* All patients are required to sign an informed consent regarding the experimental nature of this therapy, including the research biopsies, in accordance with the University of Michigan Institutional Review Board standards.
* Patients must have ECOG Performance status of 0-1.
* This study is limited to women only.
* Women of childbearing potential must have a documented negative serum HCG within 7 days prior to treatment. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

* Breast tumors that are not measurable by any of the modalities, including physical examination, mammography, or ultrasound.
* Tumors diagnosed by excisional biopsy, or incisional biopsy that does not leave measurable disease by physical examination, mammography, or ultrasound.
* Age less than 18 years.
* Granulocyte count of <1500/mm3, hemoglobin <8.0 g/dl platelet count of <100,000/mm3.
* Grade greater than or equal to 2 peripheral neuropathy.
* Hepatic

  1. Total Bilirubin > ULN
  2. AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility, as per protocol.
* Patients who are pregnant or nursing will not be eligible for this protocol.
* Patients with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil or known DPD deficiency.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months
* Any medical condition which in the opinion of the investigator puts the patient at undo risk of potentially serious complications while on this therapy.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Requirement for full dose coumadin therapy (not port prophylaxis), or a known, existing uncontrolled coagulopathy.
* Impaired renal function (estimated creatinine clearance <45ml/min as calculated with Cockcroft-Gault equation. There will be a mandated dose reduction of capecitabine for creatinine clearance < 50 ml/min to dose level -1.
* Patients must not have received any prior chemotherapy or radiation therapy for their current breast cancer. Patients who received less than 4 weeks of hormonal therapy for the treatment of the current breast cancer may be included if they agree to stop the hormonal therapy during chemotherapy. Patients who received tamoxifen or other agents for prevention of breast cancer may be included.
* Patients with active systemic malignancy in the past year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2003-07; Primary Completion 2005-05 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
specific key measurements | refer to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States